CLINICAL TRIAL: NCT00250419
Title: A Phase I Study to Evaluate the Safety/Tolerability and Immunogenicity of V-930 in Patients With Cancers Expressing HER-2 and/or CEA
Brief Title: V930 First in Man (FIM) Study (V930-002)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V930-002; 2005_047
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Cancers Expressing HER-2 and/or CEA

INTERVENTIONS:
Biological: V930

SUMMARY:
To determine the safety/tolerability, and immunogenicity of an experimental vaccine given as intramuscular injections followed by electrostimulation in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stages II, III, or IV breast, colorectal, ovaria, of non-small cell lung cancer
* Patients will either be disease free following primary therapy or have advanced disease with a durable response (>3 months) after standard therapy
* Tumor antigen HER-2 and/or CEA must be measurable in the blood or detected by Immunohistochemistry staining of the biopsies obtained from the primary tumor or metastasis

Exclusion Criteria:

* Patients with prior treatment with any HER-2 and/or CEA containing vaccine
* Patients who have significant cardiac disease
* Patients with autoimmune disorders
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Diaz CM, Chiappori A, Aurisicchio L, Bagchi A, Clark J, Dubey S, Fridman A, Fabregas JC, Marshall J, Scarselli E, La Monica N, Ciliberto G, Montero AJ. Phase 1 studies of the safety and immunogenicity of electroporated HER2/CEA DNA vaccine followed by adenoviral boost immunization in patients with solid tumors. J Transl Med. 2013 Mar 8;11:62. doi: 10.1186/1479-5876-11-62. PMID 23497415